CLINICAL TRIAL: NCT04883697
Title: Retrospective Evaluation of Risk Factors for Lower Outcomes After Vitrectomy With ILM Flap
Brief Title: Retrospective Evaluation of Risk Factors for Lower Outcomes After Vitrectomy With ILM Flap Technique
Status: Completed | Type: Observational
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Prim., Prof., MBA, Vienna Institute for Research in Ocular Surgery
Other Study IDs: RAI
Record Dates: First submitted 2021-05-01; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Macular Holes
MeSH Terms: conditions — Retinal Perforations | interventions — Vitrectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: vitrectomy with ILM peeling and ILM flap technique — outcomes after vitrectomy with ILM peeling and ILM flap technique for macukar hole repair are assessed

SUMMARY:
A retrospective review of medical charts of patients having undergone vitrectomy with ILM Peeling and ILM flap technique for macular hole repair.

DETAILED DESCRIPTION:
A retrospective review of medical charts of patients having undergone vitrectomy with ILM Peeling and ILM flap technique for macular hole repair. Pre- and postoperative OCT and visual acuity in the time period up to 6 months after surgery are reviewed and possible risk factors for failed macular hole closure or lower visual acuity outcome after surgery are assessed.

ELIGIBILITY:
Inclusion Criteria:

* Vitrectomy with ILM peeling and ILM flap technique in the time period form 1.1.2015 to 31.4.2020
* Age 18 or older

Exclusion Criteria:

* Age <18

Ages: 18 Years to 105 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all patieints have undergone vitrectomy with ILM peeling and ILM flap technique in the time period form 1.1.2015 to 31.4.2020 for macular hole repair
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
visual acuity | change between visual acuity 2-6 months postoperative to baseline
  best corrected distance visual acuity
macular hole closure | 2-6 months postoperative
  closure of the macular hole assesed with OCT

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Vienna Institute for Research in Ocular Surgery, Vienna, Austria